CLINICAL TRIAL: NCT00186758
Title: A Randomized, Sham Controlled, Crossover Trial of rTMS for Bipolar Depression
Brief Title: Transcranial Magnetic Stimulation in Bipolar Depression
Acronym: TMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Queen's University, Kingston, Ontario (Other)
Responsible Party: Dr. Gary Hasey, Director, TMS Laboratory, McMaster University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TMS2092
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Bipolar Affective Disorder
Keywords: Transcranial Magnetic Stimulation; TMS
MeSH Terms: conditions — Bipolar Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1, Phase l, True or Sham (Sham Comparator): this treatment will be True or Sham (placebo) on one side of the head, phase I
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- 2, phase ll, Sham or True (Active Comparator): This treatment will be Sham(placebo)or True on the other side of the head phase II.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Phase l clients receive either True or Sham TMS treatments on left or right side of head for 10 days.
  Phase ll clients will receive either Sham or True TMS treatments on the other side of the head - the same type as in phase l -
  Other Names: HamD; BDI II; VAS

SUMMARY:
To compare antidepressant efficacy of left or right to sham Repetitive Transcranial Magnetic Stimulation (rTMS)

to determine if non-responders can become responders if treated on the other side of the hemisphere

(rTMS)

DETAILED DESCRIPTION:
Patients will be assigned to one of 3 treatment arms for 10 days of treatment with either left high frequency or right high frequency, or sham rTMS. After 10 days of treatment, and no improvement, another 10 days of treatment follows, this time with the coil placed on the other hemisphere. Subjects will be followed for 2 months respectively with unrestricted treatment provided by their regular physician. Mood stabilizers will be continued throughout this trial.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar Depression
* no physical health problems

Exclusion Criteria:

* Metal in head/neck or skull
* History of Epilepsy
* Pregnancy
* Pacemaker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2002-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To compare antidepressant efficacy of right, left to sham | within 9 weeks

SECONDARY OUTCOMES:
To determine if QEEG activity correlates with antidepressant response to rTMS | within 9 weeks
To determine if non-responders can become responders if treating the opposite hemisphere | within 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gary Hasey, MD, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare, rTMS Laboratory, Mood Disorder Program, 100 West Fifth Street, Hamilton, Ontario, Canada